CLINICAL TRIAL: NCT02615756
Title: Molecular and Functional Neurobiology of Physical Exercise
Acronym: EXEBRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Academy of Finland (Other); Novo Nordisk A/S (Industry); Juho Vainio Foundation (Other); University of Turku (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19/180/2013
Record Dates: First submitted 2014-09-10; First posted 2015-11-26 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Physical Exercise Behavior (Liking/Aversion)
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
In this study, we use positron emission tomography (PET) and functional magnetic resonance imaging (fMRI) to study brain mechanisms that contribute to physical exercise-induced reward. We examine whether acute physical exercise releases endogenous opioids in the brain, and whether it modulates brain responses to viewing appetizing foods. Unraveling these mechanism are instrumental from a public health perspective, given the undisputed positive health effects of physical exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Native Finnish speaker
2. Age > 18 years
3. Western Caucasian origin

Exclusion Criteria:

1. Age < 18 or > 65
2. History or current mental disorder
3. BMI > 27 kg/m2
4. Use of drugs that influence the central nervous system, including nicotine
5. Poor compliance
6. Any chronic medical defect or injury which hinder or interfere everyday life
7. Eating disorder
8. Current or past excessive use of alcohol or substance abuse
9. Past dose of radiation from medical research such that the annual effective dose will exceed 10 mSv
10. Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results
11. Presence of any ferromagnetic objects that would make MR imaging contraindicated

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Binding of [11C]carfentanil in brain confirmed by positron emission tomography | Baseline and 20 min after physical exercise completion
  Change in binding of [11C]carfentanil in baseline and 20 min after physical exercise completion

CONTACTS AND LOCATIONS:
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No